CLINICAL TRIAL: NCT03807154
Title: SOLUS - A Randomized Controlled Two-site Trial Comparing Internet-based Cognitive Behavioral Therapy and Internet-based Interpersonal Psychotherapy
Brief Title: Guided Online Self-help for Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLUS
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Loneliness
Keywords: Loneliness; ICBT; Internet-based psychotherapy; Cognitive behavioral therapy; Interpersonal psychotherapy

STUDY DESIGN:
Intervention Model Description: Three conditions: Internet-based Cognitive behavioral therapy, Internet-based Interpersonal psychotherapy, and a wait-list during the primary treatment phase. The wait-list will be allocated to the two active conditions once the primary treatment phase has finished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet-based cognitive behavioral therapy (ICBT) (Experimental): A nine-week long ICBT intervention with therapist support.
  Interventions: Behavioral: ICBT
- Internet-based Interpersonal Therapy (IIPT) (Experimental): A nine-week long intervention based in interpersonal psychotherapy with therapist support.
  Interventions: Behavioral: IPT
- Wait-list (No Intervention): Wait-list control group

INTERVENTIONS:
Behavioral: ICBT — A nine week long ICBT-programme with therapist guidance. Based on cognitive and behavioral techniques that have been tailored to address loneliness.
  Arms: Internet-based cognitive behavioral therapy (ICBT)
Behavioral: IPT — A nine week long internet-based IPT-programme with therapist guidance. Contains three distinct phases: assessment phase (three weeks), focus phase (five weeks, during which the participants will choose from one of four primary problem areas during the three latter weeks), and end phase (one week).
  Arms: Internet-based Interpersonal Therapy (IIPT)

SUMMARY:
The study seeks to investigate the efficacy of two internet-based self-help programmes administered with support from a therapist. The two active conditions consist of an internet cognitive behavioral therapy (ICBT) programme and a intervention of internet-based interpersonal psychotherapy (IIPT), both of which have been developed for the present study. The active conditions will be compared to a wait-list control group.

Participants will be recruited in Sweden with a nationwide recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Frequent and distressing experiences of loneliness
* Can speak, write, and read the primary language of the country in which they reside (Sweden or the United Kingdom).
* Have access to an internet connection and a computer/smart phone/tablet
* Are prepared to participate in the study, regardless of the type of treatment they are randomly assigned to.

Exclusion Criteria:

* Changes in dosage of psychopharmaceutic medication in the last three months prior to the start of the study or a planned change during the initial treatment period.
* Other ongoing psychotherapeutic treatment
* Suicidal plans
* A previously diagnosed personality syndrome
* Ongoing substance abuse
* Other acute treatment need related to a psychiatric disorder requiring attention from a mental health professional (e.g. eating disorders such as anorexia nervosa).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Change on UCLA Loneliness Scale, Version 3 (UCLA-LS-3) | During week 2, 4, 6, and 8 of the intervention, 10 weeks after start of intervention, 4 months after completion of intervention, 12 months after start of intervention.
  Measure of loneliness, total score ranging from 20-80 (representing the sum of each of the 20 individual items). Lower scores represent less loneliness and a more favourable outcome.

SECONDARY OUTCOMES:
Change on Brunnsviken Brief Quality of Life Scale (BBQ) | 10 weeks after start of intervention, at 4 month follow-up, 12 month follow-up
  Measure of quality of life, total score ranging from 0 to 96 with a higher score indicating a higher quality of life. The scores of each of the six primary questions regarding perceived quality of life within an area of life are multiplied with the score of an item measuring the perceived importance of the area in question.
Change on Patient Health Questionnaire (PHQ-9) | 10 weeks after start of intervention, at 4 month follow-up, at 12 month follow-up
  Measure of depressive symptoms. Possible range for the total sum: 0 to 27 (created by summing up the score from each item). Clinical cut-offs for mild, moderate, moderately severe and severe major depressive disorder are considered to be 5, 10, 15, and 20 points.
Change on Social Interaction Anxiety Scale (SIAS) | 10 weeks after start of intervention, at 4 month follow-up, at 12 month follow-up
  Measure of social interaction anxiety, closely correlated with social anxiety disorder. The score on each of the 20 items are summed up. Possible range for the total sum between 0 and 80. Higher scores indicate a higher degree of social interaction anxiety.
Change on Generalised Anxiety Disorder 7-item scale (GAD-7) | 10 weeks after start of intervention, at 4 month follow-up, at 12 month follow-up
  Measure of symptoms of generalised anxiety disorder (GAD). Seven items, the score is interpreted by summing up the score from each individual item. Higher scores indicate more severe problems with worry and generalised anxiety. The total sum ranges from 0 to 21 with cut-offs of 5, 10, and 15 representing mild, moderate and severe generalised anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kall A, Back M, Welin C, Aman H, Bjerkander R, Wanman M, Lindegaard T, Berg M, Moche H, Shafran R, Andersson G. Therapist-Guided Internet-Based Treatments for Loneliness: A Randomized Controlled Three-Arm Trial Comparing Cognitive Behavioral Therapy and Interpersonal Psychotherapy. Psychother Psychosom. 2021;90(5):351-358. doi: 10.1159/000516989. Epub 2021 Jun 28. PMID 34182552